CLINICAL TRIAL: NCT00339521
Title: Genetic Susceptibility to Childhood Respiratory Illness in Mexico City
Brief Title: Genetic Susceptibility to Childhood Respiratory IIlness in Mexico City
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999028; OH99-E-N028
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Asthma
Keywords: Asthma; Mexico; Triads; Polymorphism; Genetic Predisposition
MeSH Terms: conditions — Asthma; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case-Parent Triad: Childhood Asthmatics (aged 4-17) are Cases; biologic parents of cases are genetic Controls.

SUMMARY:
We propose to add a collection of genetic material to a clinical trial of anti-oxidant supplementation for the amelioration of asthma in 7-12 year olds being conducted at a public pediatric hospital in Mexico City. The anti-oxidant study has been approved by the Institutional Review Board of the National Institute of Public Health in Mexico City and is scheduled to begin in September 1998. The purpose of this add-on study is to examine genetic polymorphisms that may be related to asthma. Asthma cases will be compared with their parents as controls. In partaicular, we will save the buffy coat from the blood collection being done on the asthmatic child for measurements of plasma micronutrients in the anti-oxidant trial for extraction of DNA. This part of the sample would otherwise be discarded. In addition, we will enroll the parents of the asthmatic child as controls for the child. From the parents, either a 10 ml blood sample or if they prefer, a sample of buccal cells will be collected. Although our current plan is to compare the asthmatic child to the parents using statistical methods based on the "transmission disequilibrium test" because research into various family designs for candidate gene studies is rapidly evolving and various sibling control sample strategies have been discussed, we would also like to collect a genetic sample on as many of the child's siblings as possible with priority given to those closest in age. This will enhance the future usefulness of the samples. We anticipate enrolling approximately 200 families....

DETAILED DESCRIPTION:
We propose to add a collection of genetic material to a clinical trial of anti-oxidant supplementation for the amelioration of asthma in 7-12 year olds being conducted at a public pediatric hospital in Mexico City. The anti-oxidant study has been approved by the Institutional Review Board of the National Institute of Public Health in Mexico City and is scheduled to begin in September 1998. The purpose of this add-on study is to examine genetic polymorphisms that may be related to asthma. Asthma cases will be compared with their parents as controls. In particular, we will save the buffy coat from the blood collection being done on the asthmatic child for measurements of plasma micronutrients in the anti-oxidant trial for extraction of DNA. This part of the sample would otherwise be discarded. In addition, we will enroll the parents of the asthmatic child as controls for the child. From the parents, either a 10 ml blood sample or if they prefer, a sample of buccal cells will be collected. Although our current plan is to compare the asthmatic child to the parents using statistical methods based on the "transmission disequilibrium test" because research into various family designs for candidate gene studies is rapidly evolving and various sibling control sample strategies have been discussed, we would also like to collect a genetic sample on as many of the child's siblings as possible with priority given to those closest in age. This will enhance the future usefulness of the samples. We anticipate enrolling approximately 200 families.

ELIGIBILITY:
* INCLUSION CRITERIA:

Moderate to severe asthma, ages 7-12 and residing within 5 km of a particular ambient air pollution monitoring station.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Asthmatic children registered at the allergy clinic of the Pediatric Hospital Frederico Gomez in Mexico City and their biological parents.
Sampling Method: Non-Probability Sample
Enrollment: 2362 (Actual)
Dates: Start 1999-05-15 (Actual); Primary Completion 2007-02-12 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
To create a resource to examine genetic susceptibility to asthma in Mexico City. | End of Study
  The role of asthma candidate genes in the association between ozone exposure and asthma incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie London, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico

REFERENCES:
- [Background] Sandford A, Weir T, Pare P. The genetics of asthma. Am J Respir Crit Care Med. 1996 Jun;153(6 Pt 1):1749-65. doi: 10.1164/ajrccm.153.6.8665031.
- [Background] Hopes E, McDougall C, Christie G, Dewar J, Wheatley A, Hall IP, Helms PJ. Association of glutamine 27 polymorphism of beta 2 adrenoceptor with reported childhood asthma: population based study. BMJ. 1998 Feb 28;316(7132):664. doi: 10.1136/bmj.316.7132.664. No abstract available. PMID 9522789
- [Background] Slutsky AS, Zamel N. Genetics of asthma: the University of Toronto Program. University of Toronto Genetics of Asthma Research Group. Am J Respir Crit Care Med. 1997 Oct;156(4 Pt 2):S130-2. doi: 10.1164/ajrccm.156.4.12tac-10. PMID 9351593